CLINICAL TRIAL: NCT05662761
Title: Assessment of the Relationship Between Severity of Chronic Venous Obstruction and Venous Claudication
Acronym: TIRED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Houman Jalaie, Deputy Head of the Department of Vascular & Endovascular Surgery of the University Hospital of AachenPD Dr. med Houman Jalaie, RWTH Aachen University
Other Study IDs: Universitätsklinikum Aachen
Record Dates: First submitted 2022-12-01; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Chronic Venous Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- symptomatic chronic obstruction: patients with symptomatic chronic obstruction of the femoroiliac and caval vein segments (VFC, VIE, VIC, VCI) treated with stent angioplasty.

SUMMARY:
Assessment of the Relationship between Severity of Chronic Venous Obstruction and Venous Claudication

DETAILED DESCRIPTION:
The postthrombotic syndrome (PTS) occurs in about 20-50% of patients after a deep Venous thrombosis and significantly affects the quality of life of patients. With the patency rates of 73-100% are achieved with endovascular procedures. At 58% of patient ulcer healing was achieved. Neglen et al. could a significant demonstrate an improvement in quality of life. Aim of the study: To show the influence of the increased inflow to venous Objectively review recanalization for patient symptoms and walking performance. Therefore, before and after venous interventions, to assess walking performance and pain-free Measure the walking distance of the patient on the treadmill and compare it to get a possible identifying relevant and/or significant changes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an obstruction in the femoral vein communis, V. iliaca externa, V. iliaca communis or V. cava inferior
2. Age: 18-80 years old
3. Signed informed consent form
4. Persons who are legally competent and mentally capable, to follow the instructions of the staff

Exclusion Criteria:

1. Patients under 18 years of age.
2. Patients who are unable to consent and/or not in are able to appreciate the nature, importance and scope of the study understand and give their consent in writing.
3. Persons acting by administrative or judicial order are housed in a facility
4. Patients who abuse drugs
5. Peripheral arterial disease stage IIb, III and IV -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with obstruction in the common femoral vein, external iliac vein, common iliac vein, or inferior vena cava
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
pain -free walking distance | 2022-2025
  pain-free walking distance after venous recanalization and stent implantation

SECONDARY OUTCOMES:
Stent openness rate | 2022-2025
  Stent openness rate
2 | 2022-2025
  Quality of life of the patients after venous recanalization and stent-lmpl.antption

CONTACTS AND LOCATIONS:
Overall Officials: Houman Jalaie, MD, Principal Investigator — Universitätsklinikum Aachen Klinik für Gefäßchirurgie
Locations (1):
- Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No